CLINICAL TRIAL: NCT02659800
Title: A Phase I and Pilot Study of the Effect of rhIL-7-hyFc (NT-I7) on CD4 Counts in Patients With High Grade Gliomas and Severe Treatment-related CD4 Lymphopenia After Concurrent Radiation and Temozolomide
Brief Title: Study of the Effect NT-I7 on CD4 Counts in Patients With High Grade Gliomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated [NCI decided to terminate ABTC Consortium due to NCI moving in different direction for Brain Cancer]
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); NeoImmuneTech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ABTC 1403; UM1CA137443 (NIH); IRB00073777 (Other: JHMIRB)
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Lymphopenia; Malignant Glioma
MeSH Terms: conditions — Lymphopenia; Glioma | interventions — efineptakin alfa

STUDY DESIGN:
Intervention Model Description: Dose Escalation - 3 levels - Group A Dexamethasone less/equal 0.75mg/day; Group B Dexamethasone greater/equal 4mg/day. At MTD Group A - w/outDexamethasone randomized Arm 1 placebo and Arm 2 MTD; Group B MTD w/ Dexamethasone single arm
Who Masked: Participant, Care Provider
Masking Description: Participant is blinded and partially randomized in the Pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A - Low Dexamethasone (LD) (Experimental): Patients receive single dose of NT-I7 IM. Treatment continues in the absence of disease progression or unacceptable toxicity. Dose Escalation
  Laboratory Biomarker Analysis Correlative Studies
  Interventions: Other: Laboratory Biomarker Analysis; Biological: NT-I7
- Arm B High Dexamethasone (HD) (Experimental): Patients receive single dose of NT-I7 IM. Treatment continues in the absence of disease progression or unacceptable toxicity. Dose Escalation
  Laboratory Biomarker Analysis Correlative Studies
  Interventions: Other: Laboratory Biomarker Analysis; Biological: NT-I7
- Arm A1 (LD) Control - Placebo (Experimental): Patients receive single dose Placebo IM (blinded). Patients also on Dexamethasone </=0.75mg daily Treatment continues in the absence of disease progression or unacceptable toxicity. Pilot
  Laboratory Biomarker Analysis Correlative Studies
  Interventions: Other: Laboratory Biomarker Analysis; Biological: NT-I7; Other: Placebo
- Arm A2 (LD) MTD (Experimental): Patients receive single dose MTD NT-I7 IM determined in Arm A (Blinded) . Patients also on Dexamethasone <=0.75mg daily Treatment continues in the absence of disease progression or unacceptable toxicity. Pilot
  Laboratory Biomarker Analysis Correlative Studies
  Interventions: Other: Laboratory Biomarker Analysis; Biological: NT-I7
- Arm B1 HD MTD (Experimental): Patients receive single dose MTD NT-I7 IM determined in Arm B (Blinded) . Patients also on Dexamethasone >= 4mg daily Treatment continues in the absence of disease progression or unacceptable toxicity. Pilot
  Laboratory Biomarker Analysis Correlative Studies
  Interventions: Other: Laboratory Biomarker Analysis; Biological: NT-I7

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: NT-I7 — Given IM
Other: Placebo — Given IM
  Arms: Arm A1 (LD) Control - Placebo

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) and select optimal biological doses (OBD) of the study drug NT-I7 in High Grade Glioma patients with severe lymphopenia, as well as to test the effect of NT-I7 on the CD4 counts of patients in comparison to control participants. This study has both a Phase I and Pilot component.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Phase I: To determine the MTD (Maximum Tolerated Dose) and select optimal biological doses (OBD) of NT-I7 in HGG patients with severe lymphopenia

Pilot Study: To test the effect of NT-I7 on CD4 counts compared to control

SECONDARY OBJECTIVES:

1. To evaluate the optimal biological dose of NT-I7
2. To evaluate the effect of concurrent dexamethasone
3. To evaluate the duration of effect on CD4 counts (up to 6 months)
4. To evaluate the total lymphocyte counts over time and serial T cell lymphocyte subtypes and the effect on T cell repertoire (up to 6 months)
5. To evaluate the serial cytokine levels (up to 6 months)
6. To evaluate the impact of adjuvant temozolomide on NT-I7 effects on CD4 counts
7. To evaluate anti-drug antibodies
8. To evaluate the pharmacokinetic profile of NT-I7 after intramuscular administration in this patient population
9. To evaluate the safety and toxicity of NT-I7 in patients with high grade glioma

OUTLINE: Patients are assigned to 1 of 2 groups depending on their use of dexamethasone.

GROUP A: Patients not on dexamethasone (or equivalent of an alternative corticosteroid), or on a dose lower than a physiologic dose (=< 0.75 mg daily)

GROUP B: patients who require dexamethasone (or equivalent of an alternative corticosteroid) => 4 mg daily

Patients must have been on the group assignment dose of corticosteroids for at least 5 days prior to the dose of NT-I7. Corticosteroid dose changes prior to the start of treatment are allowed as long as they do not alter patient's group assignment.

PHASE I TREATMENT PLAN

All patients (both Groups A and B) will be given a single dose of NT-I7 by intramuscular injection starting at 60 μg/kg, within one week after completing concurrent RT+TMZ and before starting adjuvant TMZ treatment, during the standard post-radiation break. Following this period, as per standard treatment, patients will go on to receive adjuvant temozolomide on Days 1-5 of 28-day cycles for 6 cycles. There should be about six weeks between the study injection and the start of adjuvant temozolomide; thus the start of adjuvant TMZ will be approximately two weeks later than the usual start, which is 4 weeks post-end of radiation. Patients who are delayed from receiving or are not able to receive adjuvant TMZ treatment may continue on study; adjuvant TMZ treatment is not a requirement for participation.

PILOT STUDY TREATMENT PLAN

GROUP A: participants will be given either a placebo (NT-I7 diluent) or one dose of NT-I7 at the Phase I Group A OBD by intramuscular injection within one week after completing concurrent RT+TMZ and before starting adjuvant TMZ treatment, during the standard post-radiation break.

GROUP B: participants will be given one dose of NT-I7 at the Phase I Group B OBD by intramuscular injection within one week after completing concurrent RT+TMZ and before starting adjuvant TMZ treatment, during the standard post-radiation break.

After completion of study treatment, patients are followed up every 2 months for 2 years and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed high grade glioma by pathology (World Health Organization [WHO] grade III and IV)

  * Patients' post-operative treatment must have included at least 80% of standard radiation and concomitant temozolomide; patients may not have received any other prior chemotherapy, immunotherapy or therapy with biologic agent (including immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, tumor infiltrating lymphocytes [TIL], lymphokine-activated killer [LAK] or gene therapy), or hormonal therapy for their brain tumor; prior Gliadel wafers are allowed; glucocorticoid therapy is allowed
  * Patients must have CD4 =< 300 cells/mm^3 in the last week (7 days) of standard radiation + temozolomide treatment (58-60 Gy radiation with temozolomide 75 mg/m2 daily during radiation)
  * Absolute neutrophil count >= 1,000/mcL
  * Platelets >= 50,000/mcL (need to confirm before administering study drug)
  * Hemoglobin >= 9 g/dL
  * Total bilirubin =< institutional upper limit of normal
  * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
  * Creatinine =< institutional upper limit of normal OR creatinine clearance >= 60 ml/min/1.73 m^2 for patients with creatinine levels above institutional normal
  * Activated partial thromboplastin time (APTT) or partial thromboplastin time (PTT) =< 1.5 x institutional upper limit of normal
  * Patients must have a Karnofsky performance status (KPS) >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
  * Patients must be able to provide written informed consent
  * Women of childbearing potential must have a negative serum pregnancy test prior to study entry; women of childbearing potential and men must agree to use two birth control methods (either two barrier methods or a barrier method plus a hormonal method) or abstinence prior to study entry and for the duration of study participation (through at least 90 days after the last study injection); should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
  * Dexamethasone dose must be provided for treatment group assignment:

    * Group A: patients not on dexamethasone or on a dose =< 0.75 mg daily (or equivalent of an alternative corticosteroid)
    * Group B: patients who require dexamethasone >= 4 mg daily (or equivalent of an alternative corticosteroid) ** Patients must have been on the group assignment dose of corticosteroids for at least 5 days prior to the dose of NT-I7; corticosteroid dose changes prior to the start of treatment are allowed as long as they do not alter patient's group assignment

Exclusion Criteria

* Patients receiving any other investigational agents are ineligible
* Patients with known hypersensitivity to NT-I7 or any component used in the vehicle/formulation are ineligible
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with NT-I7
* Patients with human immunodeficiency virus (HIV) are excluded
* Patients with a known or screening-period-determined corrected QT (QTc) interval > 450 msec and patients who require a therapy with a drug known to prolong the QT/QTc interval, are ineligible
* Patients with a history of or who currently have evidence of autoimmune disease (other than autoimmune thyroid disease managed with thyroid hormone replacement or vitiligo) including: myasthenia gravis, Guillain Barre syndrome, systemic lupus erythematosus, multiple sclerosis, scleroderma, ulcerative colitis, Crohn's disease, autoimmune hepatitis, Wegener's etc., are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Absolute total CD4 cell counts | At 6 weeks (after standard radiation and temozolomide treatment completion)
  The primary treatment effect is defined as an absolute increase in CD4 counts in patients treated with glycosylated recombinant human interleukin-7 compared to the control group patients without glycosylated recombinant human interleukin-7 at week 6 after radiation treatment + temozolomide treatment.

SECONDARY OUTCOMES:
Optimal dose of glycosylated recombinant human interleukin-7 determined by dose-limiting toxicities graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 | 4 weeks
  The optimal dose will be selected based on the highest absolute increase of CD4 counts compared to the control if toxicity profiles are similar between the two dose levels. Otherwise, safety will be the first consideration for dose selection. The results of the two concurrent dexamethasone groups will be summarized with standard descriptive statistics. The dose selection criteria will be similar to the non-dexamethasone groups with priority on safety rather than the highest absolute increase of CD4 counts.

CONTACTS AND LOCATIONS:
Overall Officials: Jian L Campian, MD, PhD, Study Chair — National Cancer Institute (NCI)
Locations (10):
- United States (10):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abrams Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No